CLINICAL TRIAL: NCT03797040
Title: Open-label Phase I Study to Evaluate the Safety of PLX-R18 for the Post-Exposure Prevention (PEP) or Treatment of Hematopoietic Syndrome of Acute Radiation Syndrome (HS-ARS)
Brief Title: Open-label Phase I Study for PEP or Treatment of HS-ARS PLX-R18 for the Post-Exposure Prevention (PEP) or Treatment of Hematopoietic Syndrome of Acute Radiation Syndrome (HS-ARS)
Acronym: HS-ARS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLX-R18-ARS-01
Record Dates: First submitted 2018-12-17; First posted 2019-01-08 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Ionizing Radiation Exposure
MeSH Terms: interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 4 million PLX-R18 cells/kg-up to a maximal dose of 400 million (Experimental)
  Interventions: Biological: Cell therapy

INTERVENTIONS:
Biological: Cell therapy — PLX-R18: Allogeneic ex vivo expanded placental stromal cells
  Other Names: PLX-R18

SUMMARY:
The objective of the study is to evaluate the safety of intramuscular (IM) administration of PLX-R18 in subjects exposed to ionizing radiation and who are at risk of developing HS-ARS.

Indication:Post-Exposure Prevention (PEP) or treatment of Hematopoietic Syndrome of Acute Radiation Syndrome (HS-ARS) in subjects suspected to have been exposed to ionizing radiation.

DETAILED DESCRIPTION:
This will be a Phase I, open-label safety study; each subject will receive two administrations of PLX-R18, 4 days apart. Each administration of PLX-R18 will contain 4 million cells/kg (up to a maximal dose of 400 million cells). The first administration should be preferably within 48 hours after suspected exposure and no later than 4 days after suspected exposure. The second administration will be provided 4 days after first administration.

All subjects will be hospitalized for at least 24 hours after each administration of PLX-R18,for close monitoring.In order to minimize risks, subjects will be divided in 3 sequential cohorts:

Cohort 1: 9 subjects, treated as soon as possible Cohort 2: 18 subjects, treated at least 12 hours following the first dose administered to the 9th subject Cohort 3: 33 subjects, treated at least 12 hours following the first dose administered to the 27th subject After the completion of each Cohort, stopping rules will be assessed. All subjects will receive PLX-R18 in addition to recommended care per physician discretion, based on the REMM guidelines (APPENDIX 2).

The study will be comprised of 2 periods:

Main study period - Subjects will be followed-up for 12 months and evaluated at the following time points after the first administration: Day 0 (first administration),Day 1, Day 2, Day 3, Day 4 (second administration), Day 5, Day 14 (2 weeks),Day 21 (3 weeks), Day 28 (4 weeks), Day 49 (7 weeks), Day 63 (9 weeks), Day 119(17 weeks), Day 182 (26 weeks), and Day 364 (52 weeks).Long-term survival follow-up -Week 52 to Week 260: During this period, patients will be followed-up for overall survival at: 104 weeks, 156 weeks, 208 weeks and 260 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was exposed or suspected to have been exposed to ionizing radiation of

   ≥1Gy and is at risk of developing HS-ARS, as assessed by the treating physician, based on REMM guidelines (see APPENDIX 1).
2. PLX-R18 treatment can be initiated within 4 days of exposure.
3. Aged ≥18 years.
4. Has provided informed consent. -

Exclusion Criteria:

1. Known active malignancy or history of malignancy within 3 years prior to screening except for successfully resected skin basal cell carcinoma or skin squamous cell carcinoma not located at the injection sites.
2. Known active uncontrolled infection (e.g. viral, fungal, and/or bacterial)
3. Known active infection with Hepatitis A, B, or C.
4. Pregnancy.
5. Known hypersensitivity to: Allogeneic stromal cells, dimethyl sulfoxid (DMSO), human serum albumin, or bovine products.
6. In the opinion of the Investigator the subject is at high risk of developing severe allergic/hypersensitivity reactions and a resuscitation kit including epinephrine is not at hand.
7. In the opinion of the treating physician, the subject is unsuitable for participating in the study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Any Adverse Reaction | From Week 52 to Week 260 patients will be followed-up for overall survival once a year (every 52 weeks±2 after visit 14)

SECONDARY OUTCOMES:
Recovered with no sequelae | From Week 52 to Week 260 patients will be followed-up for overall survival once a year (every 52 weeks±2 after visit 14)
  The subject has fully recovered from the AE with no residual effects observable.
Recovered with sequelae | From Week 52 to Week 260 patients will be followed-up for overall survival once a year (every 52 weeks±2 after visit 14)
  The event resolved but the subject has sequelae, which is a condition following a consequence of a disease
Ongoing AE | From Week 52 to Week 260 patients will be followed-up for overall survival once a year (every 52 weeks±2 after visit 14)
  AE is still ongoing
Overall survival | From Week 52 to Week 260 patients will be followed-up for overall survival once a year (every 52 weeks±2 after visit 14)
  Overall survival

IPD SHARING:
Plan to Share IPD: No